CLINICAL TRIAL: NCT07093827
Title: A Prospective Cohort Study on the Effect of Spinal Spinal Cord Injury on Sexual Function in Male Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Luohe Central Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: PekingUTH LXZ-SF
Record Dates: First submitted 2025-06-30; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Sexual Function Abnormal; Spinal Cord Injuries (SCI)
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Spinal Cord Injuries | interventions — Gene Fusion; Laminectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- thoracolumber fracture
  Interventions: Procedure: Posterior decompression surgery
- Cervical spinal cord injury without fracture or dislocation
  Interventions: Procedure: unilateral open-door laminoplasty
- Lumbar disc herniation
  Interventions: Procedure: Posterior lumbar discectomy with fusion
- Spine tumors
  Interventions: Procedure: Surgical resection of spinal tumors
- Ankylosing spondylitis
  Interventions: Drug: Conservative management of ankylosing spondylitis; Procedure: decompression surgery for caudal plexus disorder
- Cervical spondylosis of the spinal cord
  Interventions: Procedure: anterior cervical discectomy/fusion; Procedure: anterior cervical corpectomy/fusion
- Lumbar stenosis
  Interventions: Drug: Conservative management of lumbar spinal stenosis
- Caudal plexus disorder

INTERVENTIONS:
Procedure: Posterior decompression surgery — **Posterior decompression for thoracolumbar fractures involves a midline incision and subperiosteal exposure of the posterior spinal elements, followed by laminectomy or laminotomy to relieve neural compression. Pedicle screw-rod instrumentation is then applied above and below the fractured level under fluoroscopic guidance to restore stability, often supplemented by posterolateral fusion using bone graft. The procedure concludes with layered wound closure, providing direct neural decompression, rigid fixation for early mobilization, and reduced morbidity compared to anterior approaches in select cases. This technique is indicated for unstable fractures (e.g., AO Type B/C) or neurological deficits with posterior canal compromise, with variations based on fracture severity and surgical judgment.**
  Groups: thoracolumber fracture
Procedure: unilateral open-door laminoplasty — Posterior cervical expansive open-door laminoplasty (also known as unilateral open-door laminoplasty) is a surgical technique used to decompress the spinal cord in cervical myelopathy or spinal cord injury. The procedure involves a midline posterior cervical incision, followed by exposure of the laminae. A high-speed burr is used to create a hinged trough on one side (preserving the inner cortex) and a complete trough on the contralateral side, allowing the lamina to be gently elevated like an opening door. The opened lamina is then stabilized using sutures, miniplates, or spacers to maintain the expanded canal diameter. This approach effectively increases spinal canal space while preserving posterior elements, reducing cord compression while minimizing instability risks compared to laminectomy. It is particularly indicated for multilevel cervical stenosis with preserved cervical alignment.
  Groups: Cervical spinal cord injury without fracture or dislocation
Procedure: Posterior lumbar discectomy with fusion — Posterior lumbar discectomy with fusion (PLDF) is a standard surgical treatment for lumbar disc herniation with instability or recurrent symptoms. The procedure involves a midline posterior approach to expose the affected vertebral level, followed by laminotomy or partial laminectomy to access the neural elements. The herniated disc material is carefully removed to decompress the nerve roots, after which pedicle screws and rods are inserted for segmental stabilization. Interbody fusion (via posterior lumbar interbody fusion [PLIF] or transforaminal lumbar interbody fusion [TLIF]) is often performed by placing a bone graft or cage in the disc space to promote bony union. The combination of neural decompression, rigid instrumentation, and interbody fusion aims to relieve radicular pain while restoring spinal stability and alignment.
  Groups: Lumbar disc herniation
Procedure: Surgical resection of spinal tumors — Surgical resection of spinal tumors involves a tailored approach based on tumor location, type (primary/metastatic), and spinal stability. For posteriorly accessible lesions, a midline incision exposes the affected vertebrae, followed by laminectomy to access the epidural space and decompress neural elements. Tumor resection is performed using meticulous dissection, with intraoperative neuromonitoring to minimize neurological risk. In cases requiring vertebral body involvement, a posterolateral (costotransversectomy) or combined anterior-posterior approach may be used for en bloc or piecemeal excision. Reconstruction typically involves spinal instrumentation (pedicle screws/rods) and structural support (cages/allografts) to restore stability. The goal is maximal safe resection while preserving neurological function, often supplemented by adjuvant therapies (radiation/chemotherapy) for malignant tumors.
  Groups: Spine tumors
Drug: Conservative management of ankylosing spondylitis — Conservative management of ankylosing spondylitis (AS) focuses on symptom relief, functional preservation, and slowing disease progression through a multidisciplinary approach. First-line pharmacotherapy includes NSAIDs (e.g., celecoxib) for pain and inflammation control, supplemented by TNF-α inhibitors (e.g., adalimumab) or IL-17 inhibitors for refractory cases. Physical therapy emphasizes daily spinal extension exercises, postural training, and deep breathing to maintain mobility and prevent kyphotic deformity. Patient education on ergonomic adjustments (sleeping positions, workplace modifications) and low-impact aerobic exercise (swimming, yoga) is integral. Smoking cessation is strongly advocated due to its association with worse outcomes. Regular monitoring with inflammatory markers (CRP/ESR) and imaging (MRI for early sacroiliitis) guides therapeutic adjustments, while comorbidities (uveitis, osteoporosis) require coordinated care.
  Groups: Ankylosing spondylitis
Procedure: anterior cervical discectomy/fusion — Surgical management of cervical spondylotic myelopathy (CSM) aims to decompress the spinal cord and stabilize the spine, with the approach tailored to pathology and spinal alignment. For multilevel anterior compression, anterior cervical discectomy/fusion (ACDF) or corpectomy with plating is preferred, utilizing structural grafts or cages to restore lordosis. Posterior approaches (laminoplasty or laminectomy with fusion) are indicated for multilevel stenosis with preserved cervical curvature, employing lateral mass or pedicle screws for fixation. Hybrid strategies (e.g., ACDF combined with laminoplasty) address complex cases. Intraoperative neuromonitoring (SSEPs/MEPs) minimizes neurological risks, while emerging techniques like cervical disc arthroplasty are considered in select patients to preserve motion. Surgical timing is critical, with earlier intervention correlating to better neurological recovery in progressive myelopathy.
  Groups: Cervical spondylosis of the spinal cord
Procedure: anterior cervical corpectomy/fusion — Surgical management of cervical spondylotic myelopathy (CSM) aims to decompress the spinal cord and stabilize the spine, with the approach tailored to pathology and spinal alignment. For multilevel anterior compression, anterior cervical discectomy/fusion (ACDF) or corpectomy with plating is preferred, utilizing structural grafts or cages to restore lordosis. Posterior approaches (laminoplasty or laminectomy with fusion) are indicated for multilevel stenosis with preserved cervical curvature, employing lateral mass or pedicle screws for fixation. Hybrid strategies (e.g., ACDF combined with laminoplasty) address complex cases. Intraoperative neuromonitoring (SSEPs/MEPs) minimizes neurological risks, while emerging techniques like cervical disc arthroplasty are considered in select patients to preserve motion. Surgical timing is critical, with earlier intervention correlating to better neurological recovery in progressive myelopathy.
  Groups: Cervical spondylosis of the spinal cord
Drug: Conservative management of lumbar spinal stenosis — Conservative management of lumbar spinal stenosis (LSS) focuses on symptom alleviation and functional improvement through a multimodal approach. First-line interventions include NSAIDs or acetaminophen for neurogenic claudication pain, with consideration of epidural steroid injections for refractory radicular symptoms. Supervised physical therapy emphasizes flexion-based exercises, core stabilization, and aquatic therapy to reduce mechanical stress on neural structures. Activity modification strategies (e.g., avoiding prolonged standing) combined with assistive devices (walking frames) improve mobility. Adjuvant therapies such as gabapentinoids may be trialed for neuropathic pain, while cardiovascular conditioning (stationary cycling) counters deconditioning. Patient education on weight management and posture optimization is integral, with surgical evaluation reserved for progressive neurological deficits or failure of 3-6 months structured conservative care.
  Groups: Lumbar stenosis
Procedure: decompression surgery for caudal plexus disorder — Surgical intervention for caudal plexus disorders is indicated in cases of structural compression, trauma, or refractory symptoms unresponsive to conservative measures. The approach involves meticulous exposure of the lumbosacral plexus through a retroperitoneal or transabdominal route, depending on lesion location. For compressive pathologies, microsurgical decompression with intraoperative neurophysiological monitoring (IONM) is performed to minimize iatrogenic injury. In traumatic avulsions or sharp injuries, direct nerve repair, grafting, or neurolysis may be attempted to restore function. For chronic pain syndromes, dorsal root entry zone (DREZ) ablation or nerve decompression may be considered. Surgical success depends on etiology, timing of intervention, and extent of neural damage, with optimal outcomes achieved in early decompression of compressive lesions or precise repair of focal injuries.
  Groups: Ankylosing spondylitis

SUMMARY:
1. Background and Rationale

   Spinal cord injury (SCI) represents a devastating neurological condition with multidimensional consequences. While motor and sensory deficits are well-characterized, sexual dysfunction remains understudied despite its profound impact on quality of life. Current literature exhibits three critical gaps: (1) Limited longitudinal data on the temporal evolution of sexual dysfunction post-SCI, (2) Inadequate differentiation between psychogenic vs. neurogenic mechanisms in male patients, and (3) Heterogeneous outcome measures hindering cross-study comparisons。 This investigation builds upon pilot findings from our institution's SCI registry, where a large proportion of male participants reported clinically significant sexual impairment within 24 months post-injury. By employing standardized neuro-urological assessments alongside validated psychometric tools, this study aims to dissect the complex interplay between neurological lesion characteristics, endocrine profiles, and psychosocial adaptation processes.
2. Study Objectives

   Primary Objective To quantify the prevalence and severity trajectories of sexual dysfunction in males with SCI post-injury.

   Secondary Objectives To correlate lesion level with specific sexual function domains To identify predictors of sexual health recovery using multivariate regression modeling To establish normative data for the sexual function in SCI populations
3. Methodology

3.1 Study Design

Prospective observational cohort with three nested substudies:

Substudy A: Longitudinal biomechanical assessments Substudy B: Endocrine profiling Substudy C: Qualitative interviews exploring coping mechanisms

3.2 Participant Selection

Inclusion Criteria:

Males aged 18-60 years SCI confirmed by raiological methods or clinical symptoms Willing to participate in long-term follow-up

Exclusion Criteria:

Pre-existing sexual dysfunction History of prior surgical procedures Active psychiatric comorbidities 3.3 Data Collection Timeline Timepoint Assessments Baseline Neurological function, sexual function, raiological outcome 3-month Neurological function, sexual function, raiological outcome 12-month Neurological function, sexual function, raiological outcome 24-month Neurological function, sexual function, raiological outcome 36-month Neurological function, sexual function, raiological outcome 48-month Neurological function, sexual function, raiological outcome 60-month Neurological function, sexual function, raiological outcome

DETAILED DESCRIPTION:
Spinal cord injury (SCI) induces complex pathophysiological alterations extending beyond motor-sensory impairments, with sexual dysfunction emerging as a clinically significant yet insufficiently characterized sequela. This investigation specifically targets three critical knowledge gaps in SCI-related sexual dysfunction: First, regarding neurogenic versus psychogenic differentiation, supraspinal lesions manifest through autonomic dysreflexia-mediated hemodynamic alterations in genital perfusion, while psychological comorbidities predominantly modulate libido and arousal domains. Second, concerning temporal progression dynamics, our institutional pilot data demonstrated 68% of male SCI patients developed clinically significant sexual impairment within 24 months post-injury, though precise trajectory patterns remain uncharacterized. Third, from a biomarker integration perspective, this study will employ cortisol/DHEA-S ratio analysis combined with nocturnal penile tumescence (NPT) monitoring to objectively delineate the endocrine-neurological crosstalk underlying post-SCI sexual dysfunction pathophysiology.

This study employs a robust methodological framework comprising a primary prospective observational cohort (N=180), stratified by both anatomical lesion level and neurological impairment severity. The research architecture incorporates three integrated substudies utilizing advanced multimodal assessment protocols: Substudy A applies penile duplex ultrasonography (PDU), coupled with Rigiscan® technology, International Index of Erectile Function-5 (IIEF-5) and the Premature Ejaculation Diagnostic Tool (PEDT) to quantitatively evaluate sexual parameters; Substudy B conducts high-sensitivity LC-MS/MS serum assays (testosterone, prolactin, SHBG) to systematically characterize hypothalamic-pituitary-adrenal axis dysregulation patterns post-SCI; while Substudy C employs grounded theory methodology to analyze semi-structured interviews, establishing an evidence-based model of psychosocial coping strategy efficacy validated through the International Spinal Cord Injury Male Sexual Function (ISCI-MSF) Basic Data Set and the ICIQ-ADPHS instrument. This tripartite approach ensures comprehensive mechanistic investigation across biomechanical, endocrine, and psychosocial dimensions of post-SCI sexual dysfunction.

The study implements a comprehensive data acquisition protocol employing validated quantitative metrics across multiple domains. Longitudinal data collection occurs at predetermined intervals throughout the 60-month study period. For analytical rigor, we employ group-based trajectory modeling (GBTM) to characterize IIEF score evolution, LASSO-penalized Cox regression for time-to-recovery analysis, and partial least squares path modeling (PLS-PM) to examine mechanistic relationships between lesion level and autonomic function, endocrine profiles and arousal metrics, and depression (PHQ-9) and desire domains. Normative data development utilizes kernel density estimation to establish age-stratified IIEF reference curves, while minimum detectable change (MDC) is determined through anchor-based methods incorporating the PGIC scale, ensuring clinically meaningful interpretation of results.

This investigation incorporates several cutting-edge technical innovations to enhance methodological rigor and analytical precision: standardized biobanking procedures maintain serum aliquots to facilitate future omics-based investigations; and advanced convolutional neural networks (CNNs) automate penile duplex ultrasonography (PDU) waveform analysis to ensure objective, reproducible measurements. To maintain the highest standards of data quality, we implement robust quality assurance protocols including centralized blinding procedures for IIEF scoring (inter-rater reliability κ>0.85), multiple imputation by chained equations (MICE) to address missing data, and quarterly phantom testing of Rigiscan® equipment to verify measurement accuracy (maintaining <5% error tolerance). These integrated technological and methodological safeguards ensure the collection of high-fidelity data while enabling novel multidimensional analyses of post-SCI sexual dysfunction pathophysiology.

ELIGIBILITY:
Inclusion Criteria:

1. Biological males aged 18-60 years
2. Married or sexually active prior to injury
3. Diagnosed with pre-specified diseases
4. American Spinal Injury Association (ASIA) Impairment Scale grade B-D at admission

Exclusion Criteria:

1. Post-traumatic respiratory failure requiring mechanical ventilation
2. History of prior spinal procedures or traumatic cord injuries
3. Incomplete clinical/radiological documentation
4. Insufficient follow-up duration (<24 months post-intervention)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: A multicenter-center prospective cohort analysis of patients with pre-specified diseases treated between 2020 and 2030.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the Premature Ejaculation Diagnostic Tool (PEDT) | baseline (before injury), immediately after injury, 1, 3, 6, 12, 24, 36, 60 months after surgery
  Premature ejaculation status was determined using the PEDT, classified as confirmed (≥11, Grade 1), borderline (9-10, Grade 2), or absent (≤8, Grade 3), with lower scores reflecting improved ejaculatory control.
International Index of Erectile Function-5 (IIEF-5) | baseline (before injury), immediately after injury, 1, 3, 6, 12, 24, 36, 60 months after surgery
  Erectile function was quantitatively assessed via the IIEF-5, categorized into ordinal grades: severe dysfunction (1-7, Grade 1), moderate (8-11, Grade 2), mild (12-21, Grade 3), and normal (22-25, Grade 4), where higher scores denoted preserved erectile capacity.
American Spinal Injury Association (ASIA) Impairment Scale | baseline (before injury), immediately after injury, 1, 3, 6, 12, 24, 36, 60 months after surgery
  Neurological and functional outcomes were prospectively assessed through standardized outpatient evaluations and telemedicine follow-ups. Sensory and motor functions were classified using the ASIA Impairment Scale, the internationally recognized benchmark for spinal cord injury severity.

SECONDARY OUTCOMES:
the International Spinal Cord Injury Male Sexual Function (ISCI-MSF) Basic Data Set | immediately after injury, 1, 3, 6, 12, 24, 36, 60 months after surgery
  The ISCI-MSF Basic Data Set prospectively captured psychosexual parameters, including sexual communication willingness, reflexogenic/psychogenic erection capacity, and orgasmic function.
Torg-Pavlov ratio | immediately after injury, 1, 12, 24, 36, 60 months after surgery
  The TPR-a validated radiographic marker for developmental spinal canal stenosis-was derived by dividing mid-sagittal spinal canal diameter by corresponding vertebral body diameter on neutral lateral radiographs, measured via calibrated digital calipers.
preoperative high cord signals (HCS) in MRI T2WIs | immediately after injury, 1, 12, 24, 36, 60 months after surgery
  Intramedullary hyperintensity was quantified using mid-sagittal T2-weighted MRI: circular regions of interest (ROIs, 0.05 cm²) were delineated at sites of maximal cord hyperintensity, with reference ROIs (0.3 cm²) sampled at C7-T1 (Figure 2). The SIR was calculated as mean pathological ROI intensity divided by mean reference ROI intensity; SIR ≥1.32 defined HCS, indicative of edema, hemorrhage or liquefaction.
the rate of spinal cord compression | immediately after injury
  Spinal cord compression rate was computed from axial T2-MRI measurements as [(uncompressed anteroposterior spinal cord diameter - maximal compressed diameter)/uncompressed diameter] × 100% (Figure 3), with ≥20% denoting significant compression.
number of levels fused | immediately after surgery

OTHER OUTCOMES:
age | baseline
body mass index (BMI, kg/m²) | baseline
time interval from injury to intervention | immediately after surgery
operative duration | immediately after surgery
intraoperative blood loss | immediately after surgery
injury level(s) | immediately after injury

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided